CLINICAL TRIAL: NCT01324362
Title: A Multicenter, Randomized, Double-blind, Parallel Group, 40-week Comparison of Asthma Control Using Bronchial Hyperresponsiveness as an Additional Guide to Long-term Treatment in Adolescents and Adults Receiving Either Fluticasone Propionate/Sameterol DISKUS Twice Daily or Fluticasone Propionate DISKUS Twice Daily (or Placebo Twice Daily if Asymptomatic)
Brief Title: GSK BHR Study (Sont - Second Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM40065
Record Dates: First submitted 2011-02-03; First posted 2011-03-29 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: FP; Asthma; Sont; FSC; BHR
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Fluticasone propionate (Active Comparator)
  Interventions: Drug: Placebo; Drug: FP 100mcg; Drug: FP 250mcg; Drug: FP 500mcg
- Fluticasone propionate/salmeterol combination (Active Comparator)
  Interventions: Drug: Placebo; Drug: FSC 100/50mcg; Drug: FSC 250/50mcg; Drug: FSC500/50mcg

INTERVENTIONS:
Drug: Placebo — Twice daily dosing
  Other Names: FP 100mcg; FP 250mcg; FP 500mcg
  Arms: Fluticasone propionate
Drug: Placebo — Twice daily dosing
  Arms: Fluticasone propionate/salmeterol combination
Drug: FP 100mcg — Twice daily dosing
  Arms: Fluticasone propionate
Drug: FP 250mcg — Twice daily dosing
  Arms: Fluticasone propionate
Drug: FP 500mcg — Twice daily dosing
  Arms: Fluticasone propionate
Drug: FSC 100/50mcg — Twice daily dosing
  Arms: Fluticasone propionate/salmeterol combination
Drug: FSC 250/50mcg — Twice daily dosing
  Arms: Fluticasone propionate/salmeterol combination
Drug: FSC500/50mcg — Twice daily dosing
  Arms: Fluticasone propionate/salmeterol combination

SUMMARY:
The purpose of this study was to determine whether asthma control and reduced bronchial responsiveness could be achieved and maintained at a lower dose of inhaled corticosteroids with ADVAIR DISKUS BID or FP BID in adult and adolescent patients with persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Controller asthma medication or medium dose ICS
* Current or historical reversibility

Exclusion Criteria:

* Life-threatening asthma
* Asthma instability
* Concurrent respiratory disease
* Drug allergies
* Respiratory tract infection
* Systemic corticosteroid use
* Immunosuppressive medication use
* Postive pregnancy test
* Tobacco use
* Investigation medication use
* Site affiliation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2003-01; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Average ICS treatment dose over the treatment period | Every 8 weeks through 40 weeks of treatment

SECONDARY OUTCOMES:
Pulmonary function measures | Every 8 weeks through 40 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- United States (46):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Pueblo, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Livonia, Michigan
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Friendswood, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Brazil (3):
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
  - GSK Investigational Site, Florianópolis, Santa Catarina
  - GSK Investigational Site, São Paulo, São Paulo
- Bulgaria (2):
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- GSK Investigational Site, San Juan, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Stauffer JL, Yancey SW, Baitinger LA, Prillaman BA, Dorinsky PM. Measuring airway hyperresponsiveness: Does it add to routine measures of clinical efficacy in guiding asthma therapy? Proc Am Thorac Soc 2006;3:A213
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: SAM40065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SAM40065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAM40065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAM40065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAM40065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SAM40065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SAM40065 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register